CLINICAL TRIAL: NCT07047092
Title: Non-invasive Ventilation or CPAP in OSA-COPD Following Admission for an Acute Hypercapnic Respiratory Failure
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NOCOCA
Record Dates: First submitted 2025-06-11; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Chronic Obstructive Pulmonary Disease Exacerbation; Obstructive Sleep Apnea Exacerbation
Keywords: Chronic Obstructive Pulmonary Disease; Obstructive Sleep Apnea; Continuous Positive Airway Pressure; Non-invasive Ventilation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Sleep Apnea, Obstructive | interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant
Masking Description: Clinical experts in charge of assessing whether a hospitalization was caused by a COPD exacerbation will blinded to the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-invasive Ventilation (NIV) (Experimental): Patients randomised to the intervention arm will be established on NIV before discharge to home.
  Interventions: Device: Non-invasive Ventilation (NIV)
- Continuous Positive Airway Pressure (CPAP) (Active Comparator): Patients randomised to the control arm will be established on CPAP before discharge to home.
  Interventions: Device: Continous Positive Airway Pressure (CPAP)

INTERVENTIONS:
Device: Non-invasive Ventilation (NIV) — Patients will receive a dedicated training for the use of their NIV in the home setting. The training is the same provided in the usual care of patients established on NIV. They will choose a home care provider for the delivery of NIV as per standard care in France. A telemonitoring of adherence to NIV will be performed.
  Arms: Non-invasive Ventilation (NIV)
Device: Continous Positive Airway Pressure (CPAP) — Patients will receive a dedicated training the use of their CPAP in the home setting. The training is the same provided in the usual care of patients established on CPAP. They will choose a home care provider for the delivery of CPAP as per standard care in France. Follow-up of CPAP will be performed according to standard care in France and will therefore include a telemonitoring of adherence to CPAP.
  Arms: Continuous Positive Airway Pressure (CPAP)

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a major public health problem with 212.3 million prevalent cases of COPD worldwide and 3.3 million deaths related to COPD in 2019. Obstructive sleep apnoea (OSA) is the most common sleep disordered breathing. It is estimated that almost 1 billion adults have OSA worldwide.

Given the increasing prevalence of obesity, co-morbid OSA is frequently seen in patients with COPD. Co-morbid OSA has been shown to increase mortality, to reduce quality of life and to favour acute exacerbation of COPD. For those admitted for a life-threatening exacerbation of COPD requiring an intensive care admission for acute hypercapnic failure, they are more likely to get readmitted. For those admitted for an acute exacerbation in any ward, they are more likely to be re-admitted for another exacerbation within 180-days if their OSA is not treated.

Unfortunately, data regarding the best management of OSA in patients with co-morbid COPD are lacking as they were often excluded from clinical trials involving patients with COPD. Therefore, CPAP or NIV are administered without scientific evidence establishing which treatment is the most appropriate.

DETAILED DESCRIPTION:
Patients admitted for a severe exacerbation of COPD that required NIV or invasive ventilation or high flow therapy will be screened for the trial once they reach clinical stability that allow weaning of NIV, invasive ventilation, or high flow therapy.

The screening visit will take place during a standard consultation between 2 days following admission for acute hypercapnic respiratory failure and no later than 30 days following the discharge from the acute ward.

The inclusion visit will be performed no later than 30-days following discharge from the acute ward.

Follow-up visits will be performed at 3, 6 months after inclusion with a +/-14 days window.

Visits will be conducted in the hospital unless patient is unable to attend due to medical condition or healthcare crisis (infectious pandemic for example). In that case, a remote consultation will be performed to retrieve data available without physical attendance.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and < 85 years
2. Patient with a diagnosis of COPD according to GOLD guidelines
3. Patient admitted for an acute exacerbation of COPD requiring acute NIV or invasive ventilation or high-flow therapy (pH <7.35 with PaCO2 >45mmHg/6kPa)
4. Patient that has been weaned from acute NIV or invasive ventilation or high flow therapy
5. Patient with an overnight polygraphy or polysomnography performed 2 to 30 days following weaning from acute NIV or invasive ventilation showing an obstructive apneahypopnea index >=15/h. For patients already diagnosed with OSA, results from their prior sleep study will be retrieved. If not accessible, overnight polygraphy or polysomnography will be repeated.
6. Affiliated to the National Health Patients affiliated or, beneficiary of social security, excluding AME (Aide Médicale d'État)
7. Patient who has read and understood the information letter and signed the consent form

Exclusion Criteria:

1. Patient with NIV treatment
2. Patients who decline any use of NIV or CPAP in the home setting
3. Significant psychiatric disorder or dementia that would prevent adherence to study protocol
4. Tobacco use <10 pack-year
5. Expected survival <12 months due to any condition other than COPD.
6. Patient deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision)
7. Pregnant or breastfeeding women
8. Patient already involved in an interventional research protocol that would impact the outcome measured in the current protocol.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 386 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Demonstrate the superiority of home NIV versus home CPAP for the reduction of severe exacerbation of COPD or death. | 0-12 months from inclusion
  Reduction of severe exacerbation of COPD or death, defined by the time to occurrence of (i) death from any cause or (ii) hospitalization in relation to severe exacerbation of COPD during a follow up of 12 months after randomization.

SECONDARY OUTCOMES:
Evaluate the benefit of NIV over CPAP regarding control of sleep disordered breathing | 0-12 months from inclusion
  Control of sleep disordered breathing, defined as evolution between baseline and 1 year follow-up of the following combined criteria :
  * Apnea-hypopnea index (whilst unsupported breathing at baseline and when using the treatment overnight)
  * 3% Oxygen desaturation index (whilst unsupported breathing at baseline and when using the treatment overnight)
  * Proportion of time spent with SpO2 <90% (whilst unsupported breathing at baseline and when using the treatment overnight)
  * Change in 3% Oxygen desaturation index between baseline at 3- and 6-months follow-up when using the treatment overnight
  * Proportion of time spent with SpO2 <90% at 3 months and 6 months when using the treatment overnight.
Quality of life of NIV over CPAP | At month 3
  HRQOL compared at 3 months follow-up using HRQOL questionnaires.
Quality of life of NIV over CPAP | At month 12
  HRQOL compared at 12 months follow-up using HRQOL questionnaires.
Quality of sleep of NIV over CPAP (Pittsburgh Sleep Quality Index). | From Day 1 to Day 90
  Change in quality of sleep will be assessed using quality of sleep evaluation scales (Pittsburgh Sleep Quality Index).
Quality of sleep of NIV over CPAP | From Day 1 to Day 90
  Change in quality of sleep will be assessed using quality of sleep evaluation scales (Epworth Sleepiness Scale).
Quality of sleep of NIV over CPAP (Insomnia Severity Index). | From Day 1 to Day 90
  Change in quality of sleep will be assessed using quality of sleep evaluation scales (Insomnia Severity Index).
Quality of sleep of NIV over CPAP | From Day 1 to Day 365
  Change in quality of sleep will be assessed using the difference from baseline and one-year follow-up using quality of sleep evaluation scales (Pittsburgh Sleep Quality Index).
Quality of sleep of NIV over CPAP | From Day 1 to Day 365
  Change in quality of sleep will be assessed using the difference from baseline and one-year follow-up using quality of sleep evaluation scales (Epworth Sleepiness Scale).
Quality of sleep of NIV over CPAP (Insomnia Severity Index). | From Day 1 to Day 365
  Change in quality of sleep will be assessed using the difference from baseline and one-year follow-up using quality of sleep evaluation scales (Insomnia Severity Index).
Quality of sleep of NIV over CPAP in centres that will perform overnight polysomnography | From Day 1 to Day 365
  Quality of sleep,defined by variations between day 1 and 1 year in objective measures of sleep quality in centres that will perform overnight polysomnography : proportions of light, deep and REM sleep, wake since sleep onset, awakenings, arousals, sleep efficacy, sleep efficiency.
Respiratory function benefit of NIV over CPAP | From Day 1 to Day 365
  Respiratory function defined as change in gas exchange from baseline (Pa02, PaCO2) and 1 year: Arterial blood gas (ABG) will be measured during daytime and will be performed after 30 min on room air).
Respiratory function benefit of NIV over CPAP | At month 12
  Respiratory function defined as change in Forced Expiratory Volume 1, at 1 year.
Exercise capacity benefit of NIV over CPAP | At month 3
  Exercise capacity defined as change in distance walked during a 6MWT. 6MWT will be performed at discharge and at each follow-up visit. 6MWT will be performed according to ERS guidelines.
Exercise capacity benefit of NIV over CPAP | At month 12
  Exercise capacity defined as change in distance walked during a 6MWT at 1 year. 6MWT will be performed at discharge and at each follow-up visit. 6MWT will be performed according to ERS guidelines.
Benefit of compliance and tolerance of NIV over CPAP | From Day 1 to Day 90
  Compliance of the treatment, defined as Daily use / % of day used >4hours / side effect questionnaire, assessed at each visit.
Benefit of compliance and tolerance of NIV over CPAP | From Day 1 to Day 180
  Compliance of the treatment, defined as Daily use / % of day used >4hours / side effect questionnaire, assessed at each visit.
Benefit of compliance and tolerance of NIV over CPAP | From Day 1 to Day 365
  Compliance of the treatment, defined as Daily use / % of day used >4hours / side effect questionnaire, assessed at each visit.
Benefit of NIV over CPAP regarding usefulness of CPAP/NIV data to predict COPD severe acute exacerbation. | At month 12
  Change in breathing frequency or other extractable parameters that may predict the onset of a severe exacerbation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pitié-Salpêtrière - Sleep unit, R3S Departement, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided